CLINICAL TRIAL: NCT07232485
Title: Retinal Imaging for the Assessment of Systemic Inflammation in Endometriosis
Brief Title: Retinal Imaging for Systemic Inflammation in Endometriosis
Acronym: RISE
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 25/WS/0103
Record Dates: First submitted 2025-09-01; First posted 2025-11-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Retinal imaging; Systemic inflammation
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be taken from participants. We will keep the samples until they are used up. This may be at least 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis women: Pre-menopausal women with a previous surgical or imaging diagnosis of endometriosis
- Healthy volunteers: Pre-menopausal women with no history of endometriosis or chronic pelvic pain

SUMMARY:
There is increasing evidence that examining our eyes can tell us a lot of information about our health, and systemic diseases. Our plan is to compare the images taken of the back of eyes of women who have endometriosis with those of women who don't. We want to study what eyes can reveal about endometriosis by analyzing the retinal images from a simple noninvasive eye scan, that is already being routinely used to provide immediate clinical information in other groups of patients (eg. diabetic eye screening).

DETAILED DESCRIPTION:
What this study is about Endometriosis is now understood to affect the whole body, not just the pelvis. Many individuals with endometriosis show signs of low-grade systemic inflammation. The eye offers clinicians a clear, painless window on tiny blood vessels. Modern retinal scans can measure structure and blood flow at the back of the eye within minutes. This study will test whether retinal scans can serve as a non-invasive read-out of systemic inflammation in endometriosis. If successful, this approach could support assessment and longitudinal monitoring.

What will happen in the study

This is an exploratory case-control study. Women with endometriosis and age-matched women without endometriosis will be invited for a research visit at the Queen's Medical Research Institute (QMRI), Edinburgh. All participants will undergo the following retinal imaging:

Optical Coherence Tomography (OCT): a quick scan showing retinal and choroidal layers.

OCT Angiography (OCT-A): a map of tiny retinal vessels without dye injections. Ultra-widefield (UWF) imaging (Optos): a large-field retinal image. Scans are painless, non-invasive, and similar to routine eye assessments. The eye-imaging component takes about 30-40 minutes; the entire visit lasts about 1 hour.

Participants with endometriosis will also complete a brief endometriosis-specific quality-of-life questionnaire (EHP-30) before imaging. A small blood sample (up to 40 mL) may be taken to measure C-reactive protein (CRP) and other inflammation markers immediately or in the future (with consent). Any surplus samples may be stored securely for related research. Healthy volunteers attend a single visit only. Participants with endometriosis may be invited for repeat assessments after treatment - for example, 3 - 6 months after surgery or initiation of new hormonal therapy, or 4 - 8 weeks after completing an endometriosis-related clinical trial - to repeat the same assessments.

Burden, risks, and discomforts Retinal imaging does not use ionising radiation and is considered low risk. Possible short-lived effects include eye strain or mild headache from fixation on a target light. Venepuncture may cause brief discomfort or mild bruising. Breaks will be scheduled if needed, and expected effects will be recorded in the study file.

Measurements and analyses Scan-derived measurements will include retinal thickness, retinal nerve fibre layer thickness, macular volume, choroidal thickness, and retinal micro-vessel features. Between-group differences (endometriosis vs controls) will be analysed. Associations with blood inflammation markers will be assessed, and changes after treatment will be evaluated.

Data handling and confidentiality Study data are recorded in a case report form and entered into a secure REDCap database hosted by the University of Edinburgh. Personal details (e.g., contact information) are stored separately on secure systems with restricted access. Research data are pseudonymised using study ID codes. Data are retained and archived according to University/NHS Sponsor policies and UK data-protection law. Selected anonymised data and samples may be shared with academic or industry partners as described in the consent documents. Participation is voluntary, and participants may withdraw at any time; data collected up to withdrawal are retained for scientific and regulatory integrity.

Oversight and approvals The study is co-sponsored by the University of Edinburgh and NHS Lothian (ACCORD) and conducted in line with Good Clinical Practice (GCP) and all required approvals. Monitoring or audit may occur according to Sponsor procedures. The study ends after the last participant's last visit; a summary will be provided to the Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a previous surgical or imaging diagnosis of endometriosis

   * Pre-menopausal women and those assigned female at birth
   * Aged 18 years and over
   * A past surgical or imaging diagnosis of endometriosis within the last 5 years from date of consent
   * Ability to understand and willingness to sign the informed consent form
2. Healthy volunteers

   * Women and those assigned female at birth
   * Aged 18 years and over
   * No history of endometriosis or chronic pelvic pain
   * Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

1. Participants with a previous surgical or imaging diagnosis of endometriosis

   * The subject has donated blood (450 ml) within the last 4 weeks
   * Known reproductive tract malignancy
   * Ocular Diseases:

     * Subjects with clinically diagnosed glaucoma, optic neuropathy, optic neuritis, cataracts, or other conditions that affect the ocular structures.
     * Subjects with age-related macular degeneration, retinal vascular diseases, or other retinal disorders.
     * Subjects with any other ocular conditions that may influence the retinal or optic nerve structure.
   * Refractive Errors:

     * Subjects with high myopia (>6 diopters) or high hyperopia (>3 diopters).
     * Subjects with significant astigmatism (>2 dioptres) or other refractive errors.
   * Ocular Surgery History: Subjects with a history of ocular surgery, particularly involving the lens, cornea, retina, or optic nerve (e.g., laser vision correction, retinal surgeries, etc.).
   * Subjects with significant ocular trauma, corneal abnormalities, or active ocular infections that may interfere with OCT imaging.
   * Subjects with diabetes mellitus
2. Healthy volunteers

   * The subject has donated blood (450 ml) within the last 4 weeks
   * Known reproductive tract malignancy
   * A history of symptoms suggestive of endometriosis or chronic pelvic pain
   * Ocular Diseases:

     * Subjects with clinically diagnosed glaucoma, optic neuropathy, optic neuritis, cataracts, or other conditions that affect the ocular structures.
     * Subjects with age-related macular degeneration, retinal vascular diseases, or other retinal disorders.
     * Subjects with any other ocular conditions that may influence the retinal or optic nerve structure.
   * Refractive Errors:

     * Subjects with high myopia (>-6 dioptres) or high hyperopia (>+6 dioptres).
     * Subjects with significant astigmatism (>2 dioptres) or other refractive errors.
   * Ocular Surgery History: Subjects with a history of ocular surgery, particularly involving the lens, cornea, retina, or optic nerve (e.g., laser vision correction, retinal surgeries, etc.).
   * Subjects with significant ocular trauma, corneal abnormalities, or active ocular infections that may interfere with OCT imaging.
   * Subjects with diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women and those assigned female at birth
Study Population: This is a matched case-control study. We will recruit 50 women with endometriosis (case) and 50 women matched for age without endometriosis (controls).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Choroidal Thickness (Optical Coherence Tomography, Heidelberg SPECTRALIS) | Baseline
  Choroidal thickness quantified from OCT cross-sectional scans using the Heidelberg SPECTRALIS platform to compare endometriosis cases with matched controls at baseline.
  Unit of Measure: micrometers (µm).
Retinal Thickness (Optical Coherence Tomography, Heidelberg SPECTRALIS) | Baseline
  Full-thickness retinal measurements derived from OCT (Heidelberg SPECTRALIS) for between-group comparison at baseline.
  Unit of Measure: micrometers (µm).
Retinal Nerve Fiber Layer (RNFL) Thickness (Optical Coherence Tomography, Heidelberg SPECTRALIS) | Baseline
  RNFL thickness obtained on OCT for baseline comparison between endometriosis and matched controls.
  Unit of Measure: micrometers (µm).
Macular Volume (Optical Coherence Tomography, Heidelberg SPECTRALIS) | Baseline
  Macular volume derived from OCT volume scans for baseline between-group comparison.
  Unit of Measure: cubic millimeters (mm³).
Retinal Vessel Density (Optical Coherence Tomography Angiography, Heidelberg SPECTRALIS) | Baseline
  OCT-A-based vessel density (non-invasive angiography) used to characterize retinal microvasculature for baseline between-group comparison.
  Unit of Measure: percent (%).

SECONDARY OUTCOMES:
Change from Baseline in Choroidal Thickness | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Within-participant change from baseline to the relevant post-intervention time point(s).
  Unit of Measure: micrometers (µm).
Change from Baseline in Retinal Thickness | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Within-participant change from baseline to post-intervention. Unit of Measure: micrometers (µm).
Change from Baseline in RNFL Thickness | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Description: Within-participant change from baseline to post-intervention. Unit of Measure: micrometers (µm).
Change from Baseline in Macular Volume | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Within-participant change from baseline to post-intervention. Unit of Measure: cubic millimeters (mm³).
Change from Baseline in Retinal Vessel Density | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Within-participant change from baseline to post-intervention using OCT-A vessel density.
  Unit of Measure: percent (%).
Correlation Between Serum C-reactive Protein and Choroidal Thickness (OCT) | Baseline and post intervention (3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline)
  Association between serum CRP concentration (laboratory assay, mg/L) and choroidal thickness (OCT, µm). Pearson or Spearman as appropriate per analysis plan.
  Unit of Measure: correlation coefficient r (unitless).
Correlation Between Serum C-reactive Protein and Retinal Thickness (OCT) | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Association between serum CRP (mg/L) and retinal thickness (µm). Unit of Measure: correlation coefficient r (unitless).
Correlation Between Serum C-reactive Protein and RNFL Thickness (OCT) | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Association between serum CRP (mg/L) and RNFL thickness (µm). Unit of Measure: correlation coefficient r (unitless).
Correlation Between Serum C-reactive Protein and Macular Volume (OCT) | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Association between serum CRP (mg/L) and macular volume (mm³). Unit of Measure: correlation coefficient r (unitless).
Correlation Between Serum C-reactive Protein and Retinal Vessel Density (OCT Angiography) | Baseline; and post-intervention at 3-6 months after surgery or new hormonal treatment; or 4-8 weeks after completion of an endometriosis-related clinical trial; assessments occur within up to 3 years of baseline.
  Association between serum CRP (mg/L) and retinal vessel density (%) from OCT-A. Unit of Measure: correlation coefficient r (unitless).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Horne, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
What IPD: De-identified participant-level datasets and surplus biological samples as applicable.
  With Whom/Conditions: Academic or industry partners, as described in the PIS/consent; no release of identifiable data; publications contain no personal data.
  How/Where: Secure transfer under data-sharing agreements; data stored in validated REDCap with controlled access.
Supporting Information: Study Protocol, ICF
Time Frame: Selected anonymised data and samples collected or generated by the study may be shared with academic or industry partners within the UK from the start of the study (expected start date: 01/10/2025). Research data will be archived and stored on secure servers hosted by The University of Edinburgh (in Data Store) for 10 years.
Access Criteria: Who can access: Authorized study team and Co-Sponsor (University of Edinburgh/NHS Lothian) for conduct/monitoring/audit/archiving; Research Ethics Committee and regulators may inspect records. External academic/industry collaborators may receive selected anonymised participant-level data and anonymised surplus samples per PIS/consent; identifiable data are not released.
  What: De-identified eCRF data (demographics, clinical characteristics, retinal imaging metrics, questionnaire scores, lab reports) and, where applicable, anonymised surplus biosamples.
  How: Internal data stored in validated REDCap on secure University servers with user authentication; personal identifiers held separately; participants assigned unique study IDs (pseudonymised). External sharing only in anonymised form, under Sponsor approval and data-sharing agreements, with secure transfer. Data controller: Co-Sponsor; retention: ≥5 years for personal data, 10 years for research data.